CLINICAL TRIAL: NCT00798798
Title: Effect of Externally Implantable Tissue Expansion Device on Scar Length
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Inability to recruit eligible subjects
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, MD, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: MA-STU2545
Record Dates: First submitted 2008-11-24; First posted 2008-11-26 (Estimated); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: Skin Lesion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Implantable Tissue Expansion Device (Experimental): Will apply externally implantable tissue expansion device for 2 days
  Interventions: Device: Externally Implantable Tissue Expansion Device

INTERVENTIONS:
Device: Externally Implantable Tissue Expansion Device — Will Apply Externally Implantable Tissue Expansion Device for 2 Days

SUMMARY:
The purpose of this study is to assess whether brief use of an externally implantable tissue expansion device following excisional skin cancer surgery will significantly reduce the diameter of the final wound defect, and hence the length of the final linear primary closure. The secondary objective is to assess the functional benefits, if any, associated with use of the tissue expander.

ELIGIBILITY:
Inclusion Criteria

* Subjects ages 18-80 years old
* Subjects who are undergoing an excision of a large cutaneous lesion
* Subjects with an immediate post-excision wound defect at least 2.5 cm in diameter
* Subjects undergoing surgery on the trunk or extremities
* The subject has willingness and the ability to understand and provide informed consent for the use of their tissue and communicate with the investigator.
* Subjects who are willing to undergo no other treatments for the scars for the duration of the study.

Exclusion Criteria

* Subjects with scalp wounds
* Subjects who are unable to understand the protocol or give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-04; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Surface area (in cm2) of subject's scar | 3 months

SECONDARY OUTCOMES:
Treating physicians will note any adverse effects | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Dermatology, Chicago, Illinois, United States